CLINICAL TRIAL: NCT05776459
Title: Phase II, Multi-Center, Randomized, Blinded Study Evaluating the Efficacy, Safety and Tolerability of a Single Intratympanic Dose of AC102 Compared to Oral Steroids for the Treatment of Idiopathic Sudden Sensorineural Hearing Loss
Brief Title: Efficacy and Safety of AC102 Compared to Steroids in Adults With Idiopathic Sudden Sensorineural Hearing Loss (ISSNHL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AudioCure Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC102-201
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Hearing Loss; Hearing impairment; Hearing Loss, Sensorineural; Ear Diseases; Otorhinolaryngologic Diseases; Hearing Loss, Unilateral; Intratympanic Administration; Restoration of Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Ear Diseases; Otorhinolaryngologic Diseases; Hearing Loss, Unilateral | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AC102 (Experimental): AC102 gel and placebo tablets
  Interventions: Drug: AC102 gel; Other: Placebo Tablets
- Prednisolone (Active Comparator): Placebo gel and prednisolone tablets
  Interventions: Drug: Prednisolone; Other: Placebo gel

INTERVENTIONS:
Drug: AC102 gel — Drug: AC102 Single intratympanic injection
  Arms: AC102
Drug: Prednisolone — Active comparator: Prednisolone Tablets taken daily by mouth
  Arms: Prednisolone
Other: Placebo Tablets — Placebo Tablets taken daily by mouth
  Arms: AC102
Other: Placebo gel — Placebo Single intratympanic injection
  Arms: Prednisolone

SUMMARY:
The purpose of this Phase 2 clinical trial is to evaluate the safety, tolerability and efficacy of AC102 administered as single intratympanic injection compared to oral steroid treatment in patients with Idiopathic Sudden Sensorineural Hearing Loss (ISSNHL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 85 years
* Unilateral ISSNHL
* Onset of unilateral ISSNHL between 24 to 120 hours prior to randomization
* An absolute air conduction hearing threshold of at least 65 dB,
* Patients with a relative hearing loss of at least 30 dB compared to the current audiogram of the non-affected ear

Exclusion Criteria:

* Insufficient handling of the language used in the speech audiometry tests
* Bilateral hearing loss
* Acute hearing loss from noise trauma, barotrauma or head trauma in either ear at any time
* Congenital hearing loss
* Conductive hearing loss or combined hearing loss determined by a 4PTA > 10 dB
* History of ISSNHL in the past 1 years in the affected ear

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in pure tone audiometry (PTA; dB) | 28 days
  Mean change in absolute hearing thresholds measured by PTA from baseline to Day 28

SECONDARY OUTCOMES:
Absolute improvement of speech recognition measured in quiet compared to baseline using standardized word lists | 14, 28, 56, 84 days
  Scores between 0% to 100% correctly understood words at predefined sound pressure levels are determined

CONTACTS AND LOCATIONS:
Overall Officials: Reimar Schlingensiepen, MD, Study Director — AudioCure Pharma GmbH
Locations (39):
- Austria (4):
  - Universitätsklinik für Hals-, Nasen- und Ohrenheilkunde, Graz
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Universitätsklinik für Hals-Nasen-Ohren-Krankheiten, Salzburg
  - Universitätsklinik für Hals-, Nasen- und Ohrenkrankheiten, Vienna
- Czechia (3):
  - Zdravotnická zařízení Olomouc, ORL, Olomouc
  - Pardubická nemocnice, Klinika ORL a chirurgie hlavy a krku, Pardubice
  - Fakultní nemocnice v Motole, Prague
- Germany (15):
  - Heilig Geist Hospital, Bensheim
  - Klinik für Hals-, Nasen-, Ohrenheilkunde - Charité Campus Benjamin Franklin - HNO Hochschulambulanz, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - University Hospital Dresden 'Carl Gustav Carus' - HNO, Dresden
  - Klinik und Poliklinik für Hals-, Nasen-, Ohrenkrankheiten, Kopf- und Halschirurgie, Greifswald
  - Universitätsklinik und Poliklinik für Hals-, Nasen-, Ohrenheilkunde, Kopf- und Halschirurgie, Halle
  - HNO-Praxis Eidelstedter Platz, Hamburg
  - Klinik für Hals-, Nasen- und Ohrenheilkunde am Universitätsklinikum, Jena
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz Hals-, Nasen-, Ohrenklinik und Poliklinik, Mainz
  - Johannes Weseling Clinic Minden, Minden
  - Klinikum rechts der Isar, München
  - Evangelisches Krankenhaus - Universitätsklinik für HNO, Oldenburg
  - Universitätsklinikum Regensburg - Klinik für HNO-Heilkunde, Regensburg
  - SRH Zentralklinikum Suhl GmbH, Suhl
  - Universitätsklinikum HNO, Würzburg
- Poland (7):
  - Centrum Medyczne Kwiatowa, Bydgoszcz
  - Centrum Medyczne MAVIT - Szpital Specjalistyczny Katowice, Katowice
  - ALL-MED Cetrum Medyczne, Lodz
  - Oddział Laryngologii, Opole
  - Kliniczny Szpital Wojewódzki Nr 1 im. Fryderyka Chopina w Rzeszowie, Rzeszów
  - Uniwersytecki Szpital Kliniczny Nr 1, Szczecin
  - Trialmed, Warsaw
- Serbia (5):
  - University Clinical Centre of Serbia, Belgrade
  - Clinical Hospital Centar "dr Dragisa Misovic-Dedinje", Belgrade
  - Military Medical Academy - ENT department, Belgrade
  - Clinical Hospital Centre Zvezdara, Belgrade
  - Clinical-Hospital Center Zemun, Belgrade
- Ukraine (5):
  - Municipal non-profit enterprise Regional Clinical Hospital of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Communal non-profit enterprise "Central city clinical hospital of Ivano-Frankivsk city council", Ivano-Frankivsk
  - Municipal non-profit enterprise Oleksandrivska clinical hospital of Kyiv of the executive body of Kyiv city council, Kyiv
  - MC Universal Clinic Oberig of Kapytal LLC, Kyiv
  - LLC Clinic of Healthy Family Astramed, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes